CLINICAL TRIAL: NCT06898411
Title: Retrospective Clinical Study to Investigate the Longevity of Long-term Single Tooth Restorations From IPS e.Max CAD and Press
Brief Title: Clinical Evaluation on the Longevity of Glass Ceramic Based Single Tooth Restorations
Status: Not yet recruiting | Type: Observational
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Other Study IDs: OTCS 350528136
Record Dates: First submitted 2025-03-13; First posted 2025-03-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Single Tooth Restoration; Longevity
Keywords: crown; inlay; onlay; glass ceramic; veneer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single tooth restoration with IPS e.max: Examination of single tooth restorations with IPS e.max after a wearing time of more than 15 years.
  Interventions: Device: Single tooth restoration with IPS e.max

INTERVENTIONS:
Device: Single tooth restoration with IPS e.max — Examination of single tooth restorations with IPS e.max after a wearing time of more than 15 years. Intraoral situation will be examined similar to a standard dental examination while single tooth restorations will be documneted by photos.

SUMMARY:
This retrospective study investigates the longevity of lithium disilicate based glass-ceramic single tooth restorations placed with IPS e.max CAD and IPS e.max Press after a wearing period of more than 15 years. The primary objective is to assess the survival rate of single tooth restorations with IPS e.max CAD and IPS e.max Press after a wearing period of at least 15 years. The secondary objectives are to assess the quality of the single tooth restorations in regard of aesthetic, functional and biological properties.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years
* Informed consent signed and understood by the subject
* Received indirect single tooth restoration (inlay, onlay, veneer or crown) within the internal clinic of Ivoclar Vivadent AG between 2006 and 2010
* Single tooth restoration was done with IPS e.max CAD or IPS e.max Press
* Able to visit the internal clinic of Ivoclar Vivadent AG in Schaan, FL.

Exclusion Criteria:

* Health status (physical and mental) does not allow participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults recieving indirect single tooth restorations (inlay, onlay, veneer or crown) within the internal clinic of Ivoclar Vivadent AG between 2006 and 2010.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Survival Rate of single tooth restorations | 15 years
  Study population recieved single tooth restorations with IPS e.max between 2006-2010. After a wearing time of more than 15 years IPS e.max single tooth restorations were examined by a dentist resulting in survival rates of IPS e.max single tooth restorations after 15 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Ivoclar Vivadent AG, Schaan, Liechtenstein